CLINICAL TRIAL: NCT05256810
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled, Single Ascending and Multiple Dose Study of the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of ALN-XDH in Healthy Adult Subjects and Adult Patients With Gout
Brief Title: A Study to Evaluate ALN-XDH in Healthy Subjects and Patients With Gout
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor elected not to continue with the study
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-XDH-001; 2021-005773-68 (EudraCT Number)
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Gout
Keywords: Serum uric acid; siRNA
MeSH Terms: conditions — Gout

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part A: ALN-XDH (Experimental): A single dose of ALN-XDH administered by subcutaneous (SC) injection.
  Interventions: Drug: ALN-XDH
- Part A: Placebo (Placebo Comparator): A single dose of placebo administered by SC injection.
  Interventions: Drug: Placebo
- Part B: ALN-XDH Single Dose (Experimental): A single dose of ALN-XDH administered by SC injection.
  Interventions: Drug: ALN-XDH
- Part B: ALN-XDH Multiple Dose (Experimental): Multiple doses of ALN-XDH administered by SC injection.
  Interventions: Drug: ALN-XDH
- Part B: Placebo (Placebo Comparator): Multiple doses of placebo administered by SC injection.
  Interventions: Drug: Placebo
- Part C: ALN-XDH (Experimental): A single dose of ALN-XDH administered by SC injection.
  Interventions: Drug: ALN-XDH
- Part C: Placebo (Placebo Comparator): A single dose of placebo administered by SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-XDH — ALN-XDH administered by SC injection
  Arms: Part A: ALN-XDH; Part B: ALN-XDH Multiple Dose; Part B: ALN-XDH Single Dose; Part C: ALN-XDH
Drug: Placebo — Placebo administered by SC injection
  Arms: Part A: Placebo; Part B: Placebo; Part C: Placebo

SUMMARY:
The purpose of this study is to:

* Part A: Evaluate the safety and tolerability of single ascending doses of ALN-XDH in healthy adult participants
* Part B: Evaluate the safety, tolerability and efficacy of ALN-XDH as monotherapy in adult patients with gout
* Part C: Evaluate the safety, tolerability and efficacy of ALN-XDH as add-on therapy in adult patients with gout

ELIGIBILITY:
Inclusion Criteria:

* Part A: has serum uric acid (sUA) level ≥4 mg/dL and ≤7 mg/dL
* Parts B and C: meets the American College of Rheumatology criteria for acute arthritis of primary gout
* Part B: has an sUA level ≥8 mg/dL while not receiving urate-lowering therapy (ULT) or following a 1-week washout period of prior ULT
* Part C: has been on a stable dose of allopurinol for gout for ≥6 weeks prior to screening
* Part C: has an sUA level ≥6 mg/dL

Exclusion Criteria:

* Parts A, B and C: Has received an investigational agent within the last 30 days
* Parts A, B and C: Has experienced or is being treated for acute gout flare(s) within 14 days prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Part A: Frequency of Adverse Events | Up to 10 months
Parts B and C: Frequency of Adverse Events | Up to 14 months
Parts B and C: Percentage of Participants with Serum Uric Acid (sUA) <6 mg/dL | Up to 12.25 months

SECONDARY OUTCOMES:
Part A: Area Under the Plasma Concentration-time Curve (AUC) for ALN-XDH and Potential Metabolites | Day 1 predose and up to 48 hours postdose
Part A: Maximum Plasma Concentration (Cmax) for ALN-XDH and Potential Metabolites | Day 1 predose and up to 48 hours postdose
Part A: Time to Maximum Plasma Concentration (tmax) for ALN-XDH and Potential Metabolites | Day 1 predose and up to 48 hours postdose
Part A: Fractional Excreted in Urine (fe) for ALN-XDH and Potential Metabolites | Day 1 predose and up to 24 hours postdose
Part A: Percent Change from Baseline in sUA | Baseline through Month 9
Parts B and C: Percentage of Participants with sUA <5 mg/dL | Up to 12.25 months
Parts B and C: Percentage Change from Baseline in sUA Level | Up to 12.25 months
Parts B and C: Plasma Concentrations of ALN-XDH and Potential Major Metabolite(s) | Day 1 and Day 85 predose and up to 4 hours postdose
Parts B and C: Frequency of Treatment-associated Gout Flares | Up to 6 months
  Treatment-associated gout flares are defined as gout flares that occur within 6 months of study drug initiation.
Parts B and C: Percent Change from Baseline in 24-hour Urine Uric Acid (uUA) | Baseline through Month 6
Parts B and C: Percent Change from Baseline in Serum Xanthine | Baseline through Month 6
Parts B and C: Percent Change from Baseline in 24-hour Urine Xanthine | Baseline through Month 6
Parts B and C: Percent Change from Baseline in Serum Hypoxanthine | Baseline through Month 6
Parts B and C: Percent Change from Baseline in 24-hour Urine Hypoxanthine | Baseline through Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (1):
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badri P, Kolachana K, Duong A, Lasko M, Nandi T, Mehrotra N, Robbie GJ. Platform Assessment of Concentration-QTc Relationship Across GalNAc-siRNA Molecules. Clin Pharmacokinet. 2025 Dec 12. doi: 10.1007/s40262-025-01606-0. Online ahead of print. PMID 41388232